CLINICAL TRIAL: NCT01014988
Title: An Open-label, Multi-center, Single Arm Study to Evaluate the Safety and Tolerability of Intravenous Zanamivir in the Treatment of Hospitalized Adult, Adolescent and Pediatric Subjects With Confirmed Influenza Infection
Brief Title: Safety Study to Assess IV Zanamivir for Treatment of Influenza Infection in Patients Who Are in Hospital
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113678
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-01

CONDITIONS: Influenza, Human
Keywords: pandemic; seasonal influenza; Influenza B virus; H1N1; zanamivir; Influenza A virus, H1N1 Subtype; Relenza; influenza; neuraminidase inhibitor
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): A single arm open-label design has been selected to achieve the primary objective of providing regulatory authorities with safety data on IV zanamivir in an expedited manner. This study design also facilitates the provision of safety data on a real-time basis, if necessary.
  Interventions: Drug: zanamivir aqueous solution

INTERVENTIONS:
Drug: zanamivir aqueous solution — Zanamivir aqueous solution 10mg/mL is a clear, colorless, single use, sterile non-preserved preparation containing 10mg of zanamivir in each milliliter, and made isotonic with sodium chloride. It is presented in 20mL clear glass vials closed with rubber stoppers. Each vial contains 200mg of zanamivir.

SUMMARY:
The purpose of this study is to determine whether zanamivir aqueous solution given by intravenous injection is safe in treating hospitalized patients with confirmed influenza infection. A single arm open-label design has been selected to achieve the primary objective of providing regulatory authorities with safety data on IV zanamivir.

DETAILED DESCRIPTION:
This study will be an open-label, Phase II, multi-center, single arm study to evaluate the safety and tolerability of IV zanamivir 600mg twice daily for 5 days in hospitalized subjects with laboratory confirmed influenza infection. The initial 5-day treatment course may be extended for up to 5 additional days if viral shedding is determined to be ongoing or if clinical symptoms warrant further treatment with IV zanamivir.

Approximately 200 subjects will be enrolled into the study (approximately 150 adult/adolescent subjects and approximately 50 pediatric subjects). Adult (>/= 18 years of age) with normal renal function will receive 600mg per dose. Pediatric (6 months to <13 years)/adolescent (>13 years to <18 years) subjects will receive an age-adjusted, weight-based dose (not to exceed the 600 mg adult dose) intended to provide comparable systemic exposures to 600mg in adults. Subjects with renal impairment will receive an adjusted dose based on calculated creatinine clearance and renal replacement modality.

Serum pharmacokinetic assessments will be performed in subjects across all age groups wherever possible. Pharmacokinetic analyses will be conducted, in real-time to the extent possible, when 4 subjects (from whom samples can be obtained) are enrolled in each of the following age cohorts: 6 months to less than 1 year; 1 to less than 2 years, and 2 to less than 6 years to determine the need for pediatric dose adjustments. PK assessments are required in the first 4 subjects enrolled in the 6 months to less than 1 year age cohort, and PK data must be analyzed and IV zanamivir dosage must be reviewed before additional subjects in this age cohort can be enrolled.

The study duration is approximately 28 days for subjects whose treatment duration is 5 days, and up to approximately 33 days for subjects whose treatment duration is extended to a maximum of 10 days. The study will consist of Pre-dose Baseline Assessments (Day 1), During Treatment Assessments (Days 1 to 5, and up to Day 10), and Follow-up Assessments on the following days: Post-Treatment +2 +5, +9, +16 and +23 Days. If the first dose of IV zanamivir is administered in the afternoon/evening of Day 1, the twice daily dosing schedule will result in one treatment day encompassing two calendar days. For subjects who have been discharged from hospital, the Post-Treatment +2, +5, +9 and +16 Days Assessments can be made by telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged greater than or equal to 6 months of age; a female is eligible to enter and participate in the study if she is:

  1. of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
  2. of child-bearing potential, has a negative pregnancy test at Baseline, and agrees to one of the following methods for avoidance of pregnancy during the study and until the Post-Treatment +23 Days Follow-up Assessment:
* Abstinence; or,
* Oral contraceptive, either combined or progestogen alone; or,
* Injectable progestogen; or,
* Implants of levonorgestrel; or,
* Estrogenic vaginal ring; or,
* Percutaneous contraceptive patches; or
* Intrauterine device (IUD) or intrauterine system (IUS) showing that the expected failure rate is less than 1% per year as stated in the IUD or IUS Product Label; or,
* Has a male partner who is sterilized; or,
* Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).
* Subjects who have confirmed influenza as determined by a positive result in a rapid test for influenza A or influenza B, or a laboratory test for influenza including influenza virus antigen test, virus culture or RT-PCR test. Subjects with negative rapid test result suspected of having influenza can be enrolled following confirmatory testing by RT-PCR, antigen test or culture.
* Hospitalized subjects with symptomatic influenza
* Subjects who are able to receive their first dose of study medication within seven days of experiencing influenza-like symptoms.
* Subjects willing and able to adhere to the procedures stated in the protocol.
* Subjects/legally acceptable representative (LAR) of minors and unconscious adults willing and able to give written informed consent to participate in the study (or included as permitted by local regulatory authorities, IRBs/IECs or local laws).
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.
* UK subjects and subjects in Spain: Subjects should be in a high dependency or intensive care setting at the time of enrollment and either have severe and progressive illness on approved influenza antivirals, or are considered unsuitable for treatment with approved influenza antivirals.
* Subjects who have severe or progressive influenza illness on approved (fully licensed) influenza antivirals, or who are considered unsuitable or inappropriate for treatment with approved influenza antivirals, or who in the opinion of the investigator may benefit from IV zanamivir therapy.

Exclusion Criteria:

* Subjects who, in the opinion of the investigator, are not likely to survive the next 48 hours beyond Baseline.
* Subjects who require concurrent therapy with another influenza antiviral drug.
* Subjects who have participated in a study using an investigational influenza antiviral drug within 30 days prior to Baseline.
* Subjects who are known or suspected to be hypersensitive to any component of the study medication.
* Subjects who meet the following criteria at Baseline:
* ALT greater than or equal to 3xULN and bilirubin greater than or equal to 2xULN or ALT greater than or equal to 5xULN
* History of cardiac disease or clinically significant arrhythmia (either on ECG or by history) which, in the opinion of the Investigator, will interfere with the safety of the individual subject.
* Child in care (CiC) as defined below:

A child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation.

The definition of a CiC can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a CiC does not include a child who is adopted or has an appointed legal guardian.

* French subjects: the French subject has participated in any study using an investigational drug during the previous 30 days.
* Females who are pregnant (positive urine or serum pregnancy test at Baseline) or are breastfeeding.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (95):
- United States (36):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (8):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Chermside, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Perth, Western Australia
  - GSK Investigational Site, Subiaco, Western Australia
- Brazil (2):
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
  - GSK Investigational Site, São Paulo, São Paulo
- Canada (6):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- France (9):
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Nancy
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Tours
- GSK Investigational Site, Shatin, Hong Kong
- Japan (5):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Yamanashi
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Trondheim
- Russia (2):
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yekaterinburg
- South Africa (7):
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Observatory
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Rondebosch
  - GSK Investigational Site, Tygerberg
  - GSK Investigational Site, Worcester
- Spain (6):
  - GSK Investigational Site, (Móstoles) Madrid
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Getafe/Madrid
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (10):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Livingston, West Lothian
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Marty FM, Man CY, van der Horst C, Francois B, Garot D, Manez R, Thamlikitkul V, Lorente JA, Alvarez-Lerma F, Brealey D, Zhao HH, Weller S, Yates PJ, Peppercorn AF. Safety and pharmacokinetics of intravenous zanamivir treatment in hospitalized adults with influenza: an open-label, multicenter, single-arm, phase II study. J Infect Dis. 2014 Feb 15;209(4):542-50. doi: 10.1093/infdis/jit467. Epub 2013 Aug 27. PMID 23983212
- See also: FDA information on Influenza (Flu) antiviral drugs and related information — http://www.fda.gov/Drugs/DrugSafety/InformationbyDrugClass/ucm100228.htm
- See also: Centers For Disease Control and Prevention seasonal flu information — http://www.cdc.gov/flu/
- Available data/document: Statistical Analysis Plan: 113678 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113678 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113678 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113678 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113678 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113678 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113678 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Male or female participants who were >=6 months of age, hospitalized with laboratory-confirmed influenza, and able to receive study drug within 7 days of influenza symptom onset were enrolled in the study.
Groups:
- Cohort 6: Adults (18 Years and Older): Participants >=18 years of age received 600 milligrams (mg) zanamivir by intravenous (IV) infusion over 30 minutes twice daily, adjusted for renal function, for 5 days. Treatment could have been extended for up to 5 additional days if viral shedding or clinical symptoms warranted further treatment.
- Cohort 1: Infants (6 Months to <1 Year of Age): Participants 6 months to <1 year of age received 14 mg per kilogram (mg/kg) zanamivir by IV infusion over 30 minutes twice daily, adjusted for renal function, for 5 days. Treatment could have been extended for up to 5 additional days if viral shedding or clinical symptoms warranted further treatment.
- Cohort 2: Children (1 to <2 Years of Age): Participants 1 year to <2 years of age received 14 mg/kg zanamivir by IV infusion over 30 minutes twice daily, adjusted for renal function, for 5 days. Treatment could have been extended for up to 5 additional days if viral shedding or clinical symptoms warranted further treatment.
- Cohort 3: Children (2 to <6 Years of Age): Participants 2 years to <6 years of age received 14 mg/kg zanamivir with a maximum dose of 600 mg by IV infusion over 30 minutes twice daily, adjusted for renal function, for 5 days. Treatment could have been extended for up to 5 additional days if viral shedding or clinical symptoms warranted further treatment.
- Cohort 4: Children (6 to <13 Years of Age): Participants 6 years to <13 years of age received 12 mg/kg zanamivir with a maximum dose of 600 mg by IV infusion over 30 minutes twice daily, adjusted for renal function, for 5 days. Treatment could have been extended for up to 5 additional days if viral shedding or clinical symptoms warranted further treatment.
- Cohort 5: Adolescents (13 to <18 Years of Age): Participants 13 to <18 years of age received 12 mg/kg zanamivir with a maximum dose of 600 mg by IV infusion over 30 minutes twice daily, adjusted for renal function, for 5 days. Treatment could have been extended for up to 5 additional days if viral shedding or clinical symptoms warranted further treatment.
Period: Overall Study
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Started | 130 | 7 | 11 | 12 | 27 | 14
Completed | 107 | 7 | 9 | 12 | 26 | 11
Not Completed | 23 | 0 | 2 | 0 | 1 | 3
Not completed — Adverse Event | 20 | 0 | 1 | 0 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 6: Adults (18 Years and Older): Participants >=18 years of age received 600 mg zanamivir by IV infusion over 30 minutes twice daily, adjusted for renal function, for 5 days. Treatment could have been extended for up to 5 additional days if viral shedding or clinical symptoms warranted further treatment.
- Total: Total of all reporting groups
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age) | Total
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.30 (16.19) | 0.76 (0.127) | 1.33 (0.220) | 3.74 (1.201) | 8.67 (1.861) | 15.36 (1.151) | 33.81 (23.796)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 1 | 4 | 4 | 9 | 6 | 80
  Male | 74 | 6 | 7 | 8 | 18 | 8 | 121
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 10 | 1 | 4 | 1 | 4 | 3 | 23
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian - East Asian Heritage | 4 | 0 | 0 | 0 | 0 | 0 | 4
  Asian - South East Asian Heritage | 10 | 0 | 0 | 0 | 0 | 0 | 10
  Asian - Japanese Heritage | 0 | 1 | 0 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White - Arabic/North African Heritage | 6 | 0 | 0 | 1 | 1 | 0 | 8
  White - White/Caucasian/European Heritage | 97 | 5 | 7 | 7 | 18 | 11 | 145
  Unknown | 2 | 0 | 0 | 0 | 1 | 0 | 3
  Mixed Race | 0 | 0 | 0 | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) Considered to be Related to Study Treatment
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. All AEs were assesed by the Investigateor as related or not related to the study treatment.
Time Frame: Up to post-treatment (PT) + 23 days
Population: Safety Population: participants who received >=1 dose of study medication.
Measure: Number; unit: Participants
Groups:
- Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years): Participants 6 months to <18 years of age received 14 mg/kg zanamivir (participants from 6 months to <6 years of age) or 12 mg/kg zanamivir (participants from 6 years to <18 years of age) with a maximum dose of 600 mg by IV infusion over 30 minutes twice daily, adjusted for renal function for 5 days. Treatment could be extended for up to 5 additional days if viral shedding or clinical symptoms warranted further treatment.
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants | 28 | 5

2. Primary Outcome: Number of Participants With Any Severe or Grade 3/4 AEs
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. AEs that occured during the study were evaluated by the Investigator and graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) table for grading the severity of adult and pediatric AEs. Grade 3=severe; Grade 4=potentially life threatening.
Time Frame: Up to post-treatment (PT) + 23 days
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants | 57 | 23

3. Primary Outcome: Number of Participants With Any Severe or Grade 3/4 Treatment-related AE
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. AEs that occured during the study were evaluated by the Investigator and graded according to the DAIDS table for grading the severity of adult and pediatric AEs. Grade 3=severe; Grade 4=potentially life threatening. All AEs were assesed by the Investigateor as related or not related to the study treatment.
Time Frame: Up to post-treatment (PT) + 23 days
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants | 16 | 2

4. Primary Outcome: Number of Participants Who Permanently Discontinued the Study Treatment Due to an AE
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Time Frame: Up to 10 days
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants | 17 | 2

5. Primary Outcome: Number of Participants Who Were Permanently Discontinued From the Study Due to an AE
Description: as for outcome 4
Time Frame: Up to post-treatment (PT) + 23 days
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants | 20 | 5

6. Primary Outcome: Number of Participants With the Indicated Clinical Chemistry Values Relative to the Normal Range at Baseline (Day 1) and Day 5
Description: Blood samples for laboratory assessments were collected at Baseline (Day [D] 1), Days 3 and 5, and on post-treatment +2 days (if hospitalized) and post-treatment +23 days. Clinical chemistry parameters included alanine aminotransferase (ALT), direct bilirubin (DB), total bilirubin (TB), and creatinine. The number of participants with values that were high (H)/normal (N)/low (L) relative to the normal range at Baseline (D 1) and D 5 for the indicated clinical chemistry parameters are summarized. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline (Day 1) and Day 5
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants
  D 1, H ALT, n=129, 71 | 48 | 21
  D 1, N ALT, n=129, 71 | 79 | 49
  D 1, L ALT, n=129, 71 | 1 | 1
  D 5, H ALT, n=102, 45 | 41 | 16
  D 5, N ALT, n=102, 45 | 60 | 27
  D 5, L ALT, n=102, 45 | 1 | 1
  D 1, H DB, n=83, 60 | 17 | 9
  D 1, N DB, n=83, 60 | 61 | 45
  D 1, L DB, n=83, 60 | 2 | 3
  D 5, H DB, n=70, 36 | 20 | 4
  D 5, N DB, n=70, 36 | 46 | 28
  D 5, L DB, n=70, 36 | 1 | 1
  D 1, H TB, n=128, 71 | 11 | 13
  D 1, N TB, n=128, 71 | 110 | 50
  D 1, L TB, n=128, 71 | 7 | 7
  D 5, H TB, n=102, 42 | 13 | 6
  D 5, N TB, n=102, 42 | 85 | 32
  D 5, L TB, n=102, 42 | 4 | 2
  D 1, H Creatinine, n=128, 71 | 27 | 6
  D 1, N Creatinine, n=128, 71 | 50 | 56
  D 1, L Creatinine, n=128, 71 | 51 | 9
  D 5, H Creatinine, n=111, 46 | 31 | 7
  D 5, N Creatinine, n=111, 46 | 46 | 34
  D 5, L Creatinine, n=111, 46 | 34 | 5

7. Primary Outcome: Number of Participants With the Indicated Hematology Values Relative to the Normal Range at Baseline (Day 1) and Day 5
Description: Blood samples for laboratory assessments were collected at Baseline (Day [D] 1), Days 3 and 5, and on post-treatment +2 days (if hospitalized) and post-treatment +23 days. Hematology parameters included hemoglobin, total neutrophils (TN), and white blood cell (WBC) count. The number of participants with values that were high (H)/normal (N)/low (L) relative to the normal range at Baseline (D 1) and D 5 for the indicated hematology parameters are summarized. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline (Day 1) and Day 5
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants
  D 1, H Hemoglobin, n=130, 71 | 0 | 1
  D 1, N Hemoglobin, n=130, 71 | 48 | 30
  D 1, L Hemoglobin, n=130, 71 | 82 | 40
  D 5, H Hemoglobin, n=114, 47 | 1 | 0
  D 5, N Hemoglobin, n=114, 47 | 25 | 16
  D 5, L Hemoglobin, n=114, 47 | 88 | 31
  D 1, H TN, n=123, 70 | 51 | 34
  D 1, N TN, n=123, 70 | 59 | 29
  D 1, L TN, n=123, 70 | 13 | 7
  D 5, H TN, n=106, 45 | 49 | 20
  D 5, N TN, n=106, 45 | 49 | 18
  D 5, L TN, n=106, 45 | 8 | 7
  D 1, H WBC Count, n=130, 71 | 29 | 9
  D 1, N WBC Count, n=130, 71 | 71 | 42
  D 1, L WBC Count, n=130, 71 | 30 | 20
  D 5, H WBC Count, n=114, 47 | 50 | 12
  D 5, N WBC Count, n=114, 47 | 49 | 30
  D 5, L WBC Count, n=114, 47 | 15 | 5

8. Primary Outcome: Number of Participants With the Indicated Treatment-emergent (TE) Grade 3/4 Clinical Chemistry Toxicities
Description: A toxicity was considered to be TE if it was greater than the Baseline grade, and if it had developed or increased post-Baseline in intensity (and prior to the last dose of investigational product). Clinical chemistry parameters included ALT, TB, and creatinine. Per the DAIDS table for grading the severity of adult and pediatric AEs, Grade 3=severe and Grade 4=potentially life threatening. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to post-treatment (PT) + 23 days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants
  ALT, Grade 3, n=128, 69 | 10 | 1
  ALT, Grade 4, n=128, 69 | 5 | 0
  TB, Grade 3, n=127, 69 | 3 | 1
  TB, Grade 4, n=127, 69 | 3 | 4
  Creatinine, Grade 3, n=129, 69 | 6 | 3
  Creatinine, Grade 4, n=129, 69 | 5 | 2

9. Primary Outcome: Number of Participants With the Indicated Treatment-emergent (TE) Grade 3/4 Hematology Toxicities
Description: A toxicity was considered to be TE if it was greater than the Baseline grade, and if it had developed or increased post-Baseline in intensity (and prior to the last dose of investigational product). The hematology parameters included hemoglobin, TN, and WBC count. Per the DAIDS table for grading the severity of adult and pediatric AEs, Grade 3=severe and Grade 4=potentially life threatening. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to post-treatment (PT) + 23 days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohorts 1-5: Pediatrics/Adolescents (6 Months to <18 Years)
Number analyzed (Participants) | 130 | 71
Participants
  Hemoglobin, Grade 3, n=129, 69 | 40 | 12
  Hemoglobin, Grade 4, n=129, 69 | 9 | 2
  TN, Grade 3, n=122, 68 | 0 | 3
  TN, Grade 4, n=122, 68 | 1 | 2
  WBC count, Grade 3, n=129, 69 | 2 | 1
  WBC count, Grade 4, n=129, 69 | 2 | 0

10. Primary Outcome: Median Heart Rate at Baseline (Day 1) and Day 5
Description: Heart rate was measured at Baseline (Day 1); Days 2, 3, 4, 5, 6, 7, 8, 9, and 10; post-treatment +2 days, +5 days, +9 days, +16 days (assessments to be done if participant remained hospitalized), and +23 days. Heart rate was assessed once daily during inpatient or outpatient follow-up visits. Heart rate values at Baseline (Day 1) and Day 5 are summarized. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X, X in the category titles).
Time Frame: Baseline (Day 1) and Day 5
Population: Safety Population
Measure: Median (Full Range); unit: Beats per minute (bpm)
Groups:
- Cohort 6: Adults (18 Years and Older); Zanamivir <=5 Days: Participants >=18 years of age received 600 mg zanamivir by IV infusion over 30 minutes twice daily, adjusted for renal function, for 5 days.
- Cohort 6: Adults (18 Years and Older); Zanamivir >5 Days: Participants >=18 years of age received 600 mg zanamivir by IV infusion over 30 minutes twice daily, adjusted for renal function, for >5 days and up to 10 days if viral shedding or clinical symptoms warranted further treatment.
Arm/Group | Cohort 6: Adults (18 Years and Older); Zanamivir <=5 Days | Cohort 6: Adults (18 Years and Older); Zanamivir >5 Days | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 87 | 43 | 7 | 11 | 12 | 27 | 14
Beats per minute (bpm)
  Day 1, n=87, 43, 7, 11, 12, 27, 14 | 93.00 [58.0 to 143.0] | 95.00 [50.0 to 140.0] | 119.0 [95 to 156] | 144.0 [121 to 195] | 115.5 [92 to 160] | 112.0 [59 to 185] | 99.0 [74 to 134]
  Day 5, n=73, 42, 7, 6, 9, 15, 10 | 87.00 [50.0 to 140.0] | 93.50 [60.0 to 134.0] | 127.0 [93 to 152] | 122.5 [98 to 146] | 112.0 [85 to 123] | 102.0 [67 to 128] | 79.5 [58 to 113]

11. Primary Outcome: Median Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Baseline (Day 1) and Day 5
Description: SBP and DBP were measured at Baseline (Day 1), Days 2, 3, 4, 5, 6, 7, 8, 9, and 10; post-treatment +2 days, +5 days, +9 days, +16 days (assessments to be done if participant remained hospitalized), and +23 days. SBP and DBP were assessed once daily during inpatient or outpatient follow-up visits. SBP and DBP values at Baseline (Day 1) and Day 5 are summarized. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X, X in the category titles).
Time Frame: Baseline (Day 1) and Day 5
Population: Safety Population
Measure: Median (Full Range); unit: Millimeters of mercury (mmHg)
Arm/Group | Cohort 6: Adults (18 Years and Older); Zanamivir <=5 Days | Cohort 6: Adults (18 Years and Older); Zanamivir >5 Days | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 87 | 43 | 7 | 11 | 12 | 27 | 14
Millimeters of mercury (mmHg)
  SBP, Day 1, n=87, 43, 7, 11, 12, 27, 14 | 126.00 [70.0 to 175.0] | 118.00 [80.0 to 180.0] | 102.0 [83 to 116] | 100.0 [77 to 144] | 105.5 [82 to 124] | 108.0 [70 to 136] | 107.0 [95 to 137]
  SBP, Day 5, n=73, 43, 7, 5, 9, 15, 10 | 128.00 [51.0 to 182.0] | 132.00 [88.0 to 220.0] | 103.0 [86 to 130] | 98.0 [87 to 120] | 117.0 [83 to 140] | 110.0 [96 to 135] | 108.5 [95 to 121]
  DBP, Day 1, n=87, 43, 7, 11, 12, 27, 14 | 68.00 [32.0 to 96.0] | 63.00 [40.0 to 97.0] | 53.0 [42 to 64] | 60.0 [39 to 78] | 58.0 [37 to 86] | 57.0 [41 to 82] | 62.0 [36 to 74]
  DBP, Day 5, n=73, 43, 7, 5, 9, 15, 10 | 70.00 [29.0 to 106.0] | 66.00 [50.0 to 100.0] | 60.0 [42 to 83] | 60.0 [45 to 73] | 67.0 [43 to 89] | 68.0 [47 to 80] | 54.5 [35 to 72]

12. Primary Outcome: Median Oxygen Saturation Measured Via Transcutaneous Oximetry (TCPO2) at Baseline (Day 1) and Day 5
Description: TCPO2 is a noninvasive test that directly measures the oxygen level of tissue beneath the skin. Because oxygen is carried to tissues by blood flow in the arteries, TCPO2 is an indirect measure of blood flow. The percent (%) oxygen saturation was measured at Baseline (Day 1), Days 2, 3, 4, 5, 6, 7, 8, 9, and 10; and post-treatment +2 days, +5 days, +9 days, +16 days (assessments to be done if participant remained hospitalized), and +23 days. Oxygen saturation was assessed once daily during inpatient follow-up visits. The median oxygen saturation values at Baseline (Day 1) and Day 5 are summarized. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X, X in the category titles).
Time Frame: Baseline (Day 1) and Day 5
Population: Safety Population
Measure: Median (Full Range); unit: Percentage of oxygen level in blood
Arm/Group | Cohort 6: Adults (18 Years and Older); Zanamivir <=5 Days | Cohort 6: Adults (18 Years and Older); Zanamivir >5 Days | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 87 | 43 | 7 | 11 | 12 | 27 | 14
Percentage of oxygen level in blood
  Day 1, n=87, 43, 7, 11, 12, 27, 14 | 97.00 [82.0 to 100.0] | 96.00 [70.0 to 100.0] | 98.0 [76 to 100] | 100.0 [93 to 100] | 98.0 [93 to 100] | 98.0 [91 to 100] | 97.5 [94 to 100]
  Day 5, n=70, 43, 7, 6, 9, 15, 9 | 97.00 [73.0 to 100.0] | 96.00 [45.0 to 100.0] | 100.0 [96 to 100] | 95.5 [85 to 100] | 97.0 [95 to 100] | 97.0 [50 to 100] | 96.0 [70 to 100]

13. Primary Outcome: Median Respiration Rate at Baseline (Day 1) and Day 5
Description: Respiration rate was measured at Baseline (Day 1), Days 2, 3, 4, 5, 6, 7, 8, 9, and 10; and post-treatment +2 days, +5 days, +9 days, +16 days (assessments to be done if participant remained hospitalized), and +23 days. Respiration rate was assessed once daily during inpatient or outpatient follow-up visits. The median respiration rate at Baseline (Day 1) and Day 5 is summarized. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X, X in the category titles).
Time Frame: Baseline (Day 1) and Day 5
Population: Safety Population
Measure: Median (Full Range); unit: Breaths per minute
Arm/Group | Cohort 6: Adults (18 Years and Older); Zanamivir <=5 Days | Cohort 6: Adults (18 Years and Older); Zanamivir >5 Days | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 87 | 43 | 7 | 11 | 12 | 27 | 14
Breaths per minute
  Day 1, n=87, 43, 7, 11, 12, 27, 14 | 23.00 [6.0 to 47.0] | 22.00 [10.0 to 40.0] | 32.0 [28 to 46] | 34.0 [20 to 40] | 29.5 [22 to 66] | 20.0 [4 to 49] | 21.0 [0 to 98]
  Day 5, n=67, 42, 7, 6, 9, 15, 10 | 20.00 [10.0 to 42.0] | 23.50 [8.0 to 41.0] | 40.0 [28 to 48] | 31.0 [10 to 50] | 30.0 [22 to 44] | 23.0 [8 to 48] | 19.0 [0 to 28]

14. Primary Outcome: Median Body Temperature at Baseline (Day 1) and Day 5
Description: Body temperature was recorded at Baseline (Day 1), Days 2, 3, 4, 5, 6, 7, 8, 9, and 10; and post-treatment +2 days, +5 days, +9 days, +16 days (assessments to be done if participant remained hospitalized), and +23 days. Body temperature was recorded once daily during inpatient or outpatient follow-up visits. Median body temperature at Baseline (Day 1) and Day 5 is summarized. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X, X in the category titles).
Time Frame: Baseline (Day 1) and Day 5
Population: Safety Population
Measure: Median (Full Range); unit: Degrees centigrade
Arm/Group | Cohort 6: Adults (18 Years and Older); Zanamivir <=5 Days | Cohort 6: Adults (18 Years and Older); Zanamivir >5 Days | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 87 | 43 | 7 | 11 | 12 | 27 | 14
Degrees centigrade
  Day 1, n=87, 43, 7, 11, 12, 27, 14 | 37.30 [33.4 to 40.1] | 37.30 [35.3 to 40.4] | 36.8 [36 to 40] | 37.3 [34 to 40] | 37.5 [36 to 39] | 37.3 [33 to 39] | 37.5 [36 to 40]
  Day 5, n=73, 42, 7, 6, 9, 15, 10 | 37.00 [35.3 to 38.8] | 37.15 [34.5 to 39.8] | 37.0 [36 to 38] | 36.8 [36 to 38] | 37.3 [37 to 38] | 37.1 [37 to 39] | 37.1 [37 to 39]

15. Primary Outcome: Number of Participants Assessed as Normal/Abnormal (Clinically Significant [CS] and Not Clinically Significant [NCS]) for 12-lead Electrocardiogram (ECG) at Baseline (Day 1)
Description: The number of participants with an ECG status of normal and abnormal CS or NCS, as determined by the Investigator, is reported. Normal=all ECG parameters within the accepted normal ranges. Abnormal=ECG findings outside of normal ranges. CS=ECG with a CS abnormality that meets exclusion criteria. NCS=ECG with an abnormality that is not CS nor meets exclusion criteria, per Investigator, based on reasonable standards of clinical judgment. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X in the category titles).
Time Frame: Baseline (Day 1)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14
Participants
  Normal, n=128, 7, 10, 12, 25, 13 | 68 | 5 | 7 | 8 | 20 | 8
  Abnormal NCS, n=128, 7, 10, 12, 25, 13 | 57 | 2 | 2 | 4 | 5 | 5
  Abnormal CS, n=128, 7, 10, 12, 25, 13 | 7 | 0 | 1 | 0 | 0 | 0

16. Primary Outcome: Median Corrected QT Interval (QTc) for Heart Rate by Fridericia's Formula (QTcF) and Bazett's Formula (QTcB) at Baseline (Day 1) and Day 5
Description: Twelve-lead ECGs were recorded for the parameters of QTcF and QTcB. The first set of pre-dose ECG values at Baseline (Day 1) and the pre-dose ECG values at Day 5 are presented. Baseline is defined as the last pre-treatment value collected. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X, X in the category titles). "NA" indicates that data are not available/analysis was not performed. Cohort 1 QTcF and QTcB minimum values of 0.0 were data entry errors that could not be addressed after Data Base Freeze.
Time Frame: Baseline (Day 1) and Day 5
Population: Safety Population
Measure: Median (Full Range); unit: Milliseconds
Arm/Group | Cohort 6: Adults (18 Years and Older); Zanamivir <=5 Days | Cohort 6: Adults (18 Years and Older); Zanamivir >5 Days | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 87 | 43 | 7 | 11 | 12 | 27 | 14
Milliseconds
  QTcF, Baseline, n=87, 42, 6, 9, 11, 24, 13 | 400.6 [204 to 584] | 413.5 [285 to 502] | 356.00 [0.0 to 465.0] | 362.00 [331.0 to 426.0] | 365.00 [297.0 to 483.0] | 387.50 [267.0 to 544.0] | 387.00 [271.0 to 424.0]
  QTcF, Day 5, n=68, 40, 0, 1, 3, 3, 5 | 406.6 [298 to 610] | 405.5 [339 to 555] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | 373.00 [373.00 to 373.00] | 394.00 [291.0 to 411.0] | 353.00 [310.0 to 392.0] | 389.00 [179.0 to 409.0]
  QTcB, Baseline, n=87, 42, 6, 9, 11, 24, 13 | 424.0 [231 to 642] | 432.0 [310 to 514] | 412.00 [0.0 to 443.0] | 422.00 [389.0 to 502.0] | 410.00 [330.0 to 493.0] | 422.50 [264.0 to 497.0] | 415.00 [316.0 to 467.0]
  QTcB, Day 5, n=68, 40, 0, 1, 3, 3, 5 | 422.0 [325 to 649] | 434.0 [334 to 535] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | 416.00 [416.0 to 416.0] | 444.00 [321.0 to 475.0] | 380.00 [350.0 to 410.0] | 399.00 [189.0 to 422.0]

17. Secondary Outcome: Median Time to Virologic Improvement
Description: Time to virologic improvement is defined as a 2-log drop in viral load or undetectable viral ribonucleic acid (RNA) as measured by quantitative reverse transcriptase-polymerase chain reaction (RT-PCR) from nasopharyngeal samples (PCR positive at Baseline). Only those participants available at the specified time points were analyzed.
Time Frame: Up to post-treatment (PT) + 23 days
Population: ITT-E Population consisted of all participants who receiveed at least one dose of IV zanamivir.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 76 | 5 | 7 | 9 | 13 | 7
Days | 3.0 [1 to 26] | 4.0 [2 to 9] | 4.0 [3 to 25] | 3.0 [3 to 7] | 5.0 [3 to 6] | 4.0 [2 to 13]

18. Secondary Outcome: Median Change From Baseline (Influenza A or B Quantitative PCR, as Appropriate) in Viral Load at the Indicated Time Points
Description: Change from Baseline in viral load was measured from nasopharyngeal swab samples, as determined by RT-PCR (PCR positive at Baseline). Nasopharyngeal swab samples were collected at Baseline (Day 1); Day 2, Day 3, Day 4, Day 5, Day 7, and Day 10; and, only if the participants had continued symptoms and were hospitalized, post-treatment (PT) samples were collected at +2 days, +5 days, +9 days, +16 days, and +23 days. 'PT +23 days' also comprises viral load values at early study withdrawal. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X in the category titles). "NA" indicates that data are not available/analysis was not performed.
Time Frame: Baseline (Day 1); Days 2, 3, 4, 5, 7, and 10; and post-treatment +2, +5, +9, +16, +23 days
Population: ITT-E Population
Measure: Median (Full Range); unit: Log10 copies per milliliter
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14
Log10 copies per milliliter
  Day 2, n=89, 0, 0, 2, 3, 2 | -0.92 [-4.00 to 2.00] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -3.750 [-3.87 to -3.63] | -1.160 [-1.87 to -0.50] | -2.280 [-2.55 to -2.01]
  Day 3, n=82, 4, 7, 10, 15, 7 | -1.42 [-3.38 to 1.08] | -1.655 [-3.15 to -0.94] | -1.930 [-4.36 to 0.55] | -2.215 [-6.16 to -0.49] | -1.330 [-5.19 to 0.62] | -2.550 [-4.01 to -0.29]
  Day 4, n=84, 0, 0, 2, 2, 1 | -1.59 [-5.40 to 1.38] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -4.895 [-5.01 to -4.78] | -2.060 [-2.60 to -1.52] | -2.550 [-2.55 to -2.55]
  Day 5, n=75, 5, 4, 8, 12, 5 | -1.57 [-5.06 to 2.05] | -2.720 [-4.92 to -0.12] | -3.705 [-6.20 to 0.24] | -3.285 [-6.16 to -1.81] | -2.930 [-6.71 to -1.53] | -2.550 [-4.01 to -1.40]
  Day 7, n=23, 1, 1, 1, 3, 1 | -1.58 [-3.52 to 3.02] | -1.820 [-1.82 to -1.82] | -6.200 [-6.20 to -6.20] | -3.030 [-3.03 to -3.03] | -3.040 [-3.46 to -1.26] | -1.610 [-1.61 to -1.61]
  Day 10, n=19, 0, 2, 1, 4, 1 | -1.75 [-4.00 to 2.04] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -5.385 [-6.20 to -4.57] | -6.430 [-6.43 to -6.43] | -4.760 [-5.42 to -2.48] | -1.670 [-1.67 to -1.67]
  PT +2 days, n=32, 0, 1, 2, 6, 3 | -1.38 [-4.86 to 0.46] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -6.200 [-6.20 to -6.20] | -2.495 [-2.91 to -2.08] | -3.825 [-5.42 to -1.60] | -3.060 [-4.61 to -1.63]
  PT +5 days, n=26, 0, 2, 0, 5, 2 | -1.84 [-5.21 to -0.40] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -5.385 [-6.20 to -4.57] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -4.190 [-5.42 to -1.60] | -3.275 [-3.43 to -3.12]
  PT +9 days, n=27, 0, 1, 0, 3, 2 | -2.58 [-5.21 to -0.41] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -6.200 [-6.20 to -6.20] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -4.190 [-5.42 to -1.60] | -3.865 [-4.61 to -3.12]
  PT +16 days, n=21, 0, 1, 0, 4, 1 | -2.48 [-5.21 to -0.41] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -2.950 [-2.95 to -2.95] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -3.825 [-4.56 to -1.60] | -4.610 [-4.61 to -4.61]
  PT +23 days, n=21, 2, 4, 0, 4, 0 | -2.89 [-5.21 to -0.46] | -4.455 [-4.92 to -3.99] | -4.670 [-6.20 to -2.95] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed. | -3.825 [-4.56 to -1.60] | NA [NA to NA] — "NA" indicates that data are not available/analysis was not performed.

19. Secondary Outcome: Mean Viral Susceptibility to Zanamivir at Baseline (Day 1) and All Post-Baseline Visits Collectively
Description: Viral susceptibility to zanamivir at Baseline and at all post-Baseline visits collectively was assessed by neuraminidase (NA) enzyme inhibition assay. The mean IC50 data are summarized by subtype (A/H1N1, A/H3N2, B) and by visit. IC50 is defined as the concentration of zanamvir required to inhibit NA activity by 50%. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). "NA" indicates that data are not available/analysis was not performed. Please note: pediatric data are pending and will be updated when available.
Time Frame: Baseline and up to post-treatment (PT) + 23 days
Population: ITT-E Population
Measure: Mean (Standard Deviation); unit: Nanomolar (nM)
Arm/Group | Cohort 6: Adults (18 Years and Older)
Number analyzed (Participants) | 130
Nanomolar (nM)
  A/H1N1, Day 1, n=22, 2 | 0.2091 (0.06886)
  A/H1N1, All Post-Baseline, n=8, 1 | 0.1800 (0.04000)
  A/H3N2, Day 1, n=5, 16 | 0.2660 (0.08385)
  A/H3N2, All Post-Baseline, n=2, 3 | 0.2300 (0.01414)
  B, Day 1, n=2, 16 | 1.6100 (0.35355)
  B, All Post-Baseline, n=0, 10 | NA (NA) — "NA" indicates that data are not available/analysis was not performed.

20. Secondary Outcome: Number of Participants With Treatment-emergent (TE) Mutations
Description: Viral RNA isolated from participants at Baseline (Day 1) and post-Baseline visits were sequenced to determine the presence of TE neuraminidase (NA) and hemagglutinin (HA) mutations resulting from selective pressure. A mutation was considered to be TE if it was not present at Baseline and was present in the last post-Baseline sample analyzed.These mutations were classified as either known to confer zanamvir resistance or novel mutations with unknown clinical significance. Please note: pediatric data are pending and will be updated when available.
Time Frame: Baseline and up to post-treatment (PT) + 23 days
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older)
Number analyzed (Participants) | 130
Participants
  Known Zanamivir-Resistant NA Mutations | 0
  Novel NA Mutations | 5
  Resistant HA Mutations | 2
  Novel HA Mutations | 4

21. Secondary Outcome: Median Time to Resolution of Individual Vital Signs
Description: Times to return to afebrile status (normal body temperature), normal respiratory status, normal heart rate, and normal systolic blood pressure were assessed. Afebrile status is defined as a temperature <=36.6 axilla, <=37.2 oral, or <=37.7 rectal, core or typanic, degrees Centigrade. A return to normal respiratory status is defined as either: (a) return to pre-morbid oxygen requirement; or (b) return to no need for supplemental oxygen; or (c) respiratory rate <=60, <=40, <=34, <=30, <=24 or <=24 breaths/minute (without supplemental oxygen) for Cohorts 1-6 respectively . A normal HR is defined as <=160, <=150, <=140, <=120, <=100 or <=100 bpm for Cohorts 1-6 respectively, and a normal SBP is defined as >=70, >=74, >=76, >=80, >=90 or >=90 mmHg for Cohorts 1-6 respectively. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X in the category titles).
Time Frame: Up to post-treatment (PT) + 23 days
Population: ITT-E Population
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14
Days
  Afebrile Status, n=120, 7, 11, 7, 24, 13 | 3.0 [2 to 34] | 4.0 [2 to 26] | 2.0 [1 to 30] | 25.0 [2 to 32] | 3.0 [2 to 26] | 3.0 [2 to 15]
  Respiratory Status, n=89, 7, 10, 12, 23, 9 | 8.0 [2 to 36] | 5.0 [2 to 16] | 2.0 [1 to 21] | 3.5 [2 to 21] | 3.0 [2 to 33] | 2.0 [2 to 20]
  HR, n=121, 7, 11, 12, 27, 13 | 2.0 [2 to 22] | 2.0 [2 to 2] | 2.0 [1 to 25] | 2.0 [2 to 3] | 2.0 [2 to 31] | 2.0 [2 to 5]
  SBP, n=128, 7, 11, 12, 27, 14 | 2.0 [2 to 3] | 2.0 [2 to 2] | 2.0 [1 to 3] | 2.0 [2 to 3] | 2.0 [2 to 24] | 2.0 [2 to 3]

22. Secondary Outcome: Number of Participants With the Indicated Ventilation Status: Modality of Supplemental Oxygen Delivery and Mechanical Ventilation
Description: Ventilation status was measured at Baseline (Day 1); Days 2, 3, 4, 5, 6, 7, 8, 9, and 10; and post-treatment +2 days, +5 days, +9 days, +16 days (assessments to be done if participant remained hospitalized), and +23 days. Ventilation status was assessed once daily during inpatient follow-up visits. The number of participants reported for machine-assisted: extracorporeal membrane oxygenation (ECMO), endotracheal mechanical ventilation, and supplemental oxygen delivery (SOD) at "any time (AT) on study" and at Baseline (Day 1) are summarized.
Time Frame: Up to post-treatment (PT) + 23 days
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14
Participants
  AT on Study, Machine-Assisted: ECMO | 4 | 0 | 1 | 0 | 2 | 1
  AT on Study, Machine-Assisted: Endotracheal | 74 | 3 | 5 | 4 | 14 | 4
  AT on Study, SOD | 91 | 3 | 5 | 7 | 13 | 5
  Day 1, Machine-Assisted: ECMO | 3 | 0 | 1 | 0 | 2 | 1
  Day 1, Machine-Assisted: Endotracheal | 60 | 2 | 3 | 4 | 11 | 4
  Day 1, SOD | 46 | 1 | 3 | 1 | 6 | 1

23. Secondary Outcome: Duration of Mechanical Ventilation and Supplemental Oxygen Use
Description: Due to the conditional nature of data collection post treatment, the duration of mechanical ventilation and supplemental oxygen use were not determined.
Time Frame: Up to discharge from the hospital
Population: ITT-E Population
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Median Time to Return to Pre-morbid Functional Status
Description: Time to return to pre-morbid functional status was assessed on a 3-point scale (bed rest, limited ambulation, or unrestricted). Only those participants available at the specified time points were analyzed.
Time Frame: Up to post-treatment (PT) + 23 days
Population: ITT-E Population
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 76 | 7 | 9 | 11 | 22 | 9
Days | 10.0 [2 to 48] | 8.0 [2 to 27] | 3.0 [2 to 27] | 5.0 [2 to 28] | 5.5 [2 to 34] | 4.0 [2 to 8]

25. Secondary Outcome: Number of Participants With the Indicated Mortality Status at Day 14 and Day 28
Description: The number of participants who died on or before Study Day 14 and Study Day 28 was summarized. Only those participants available at the specified time points were analyzed.
Time Frame: Day 14 and Day 28
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14
Participants
  Died on or before Study Day 14, No | 113 | 7 | 11 | 12 | 26 | 12
  Died on or before Study Day 14, Yes | 17 | 0 | 0 | 0 | 1 | 2
  Died on or before Study Day 28, No | 108 | 7 | 10 | 12 | 26 | 11
  Died on or before Study Day 28, Yes | 22 | 0 | 1 | 0 | 1 | 3

26. Secondary Outcome: Median Time to Clinical Response (Sustained Resolution) of All Vital Signs (Composite)
Description: Sustained resolution of the following vital signs (composite) was assessed: afebrile status, normal oxygen saturation, normal respiratory status, normal HR, and normal BP. Clinical response is defined as the resolution of at least four of five vital signs within the following resolution criteria, maintained for 24 hours or hospital discharge, whichever occurred first: Temperature in degrees Centigrade (<=36.6 axilla, <=37.2 oral, <=37.7 rectal, core or tympanic); oxygen saturation (>=95%, without supplemental oxygen); respiratory status (return to pre-morbid oxygen requirement, or no need for supplemental oxygen, or respiratory rate <=60, <=40, <=34, <=30, <=24 or <=24 breaths/minute without supplemental oxygen for Cohorts 1-6 respectively); HR (<=160, <=150, <=140, <=120, <=100 or <=100 bpm for Cohorts 1-6 respectively); SBP (>=70, >=74, >=76, >=80, >=90 or >=90 mmHg for Cohorts 1-6 respectively). Only those participants available at the specified time points were analyzed.
Time Frame: Up to post-treatment (PT) + 23 days
Population: ITT-E Population
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 81 | 7 | 10 | 12 | 25 | 11
Days | 9.0 [2 to 32] | 7.0 [2 to 23] | 3.5 [1 to 21] | 6.5 [2 to 37] | 4.0 [1 to 42] | 5.0 [2 to 32]

27. Secondary Outcome: Number of Participants With Any AE Categorized as an Influenza Complication
Description: as for outcome 4
Time Frame: Up to post-treatment (PT) + 23 days
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14
Participants | 45 | 4 | 4 | 3 | 8 | 3

28. Secondary Outcome: Number of Participants Who Used Any Concomitant Antibiotic Medications for Complications of Influenza
Description: Concomitant medications (prescription and non-prescription) were permitted during the course of the study at the Investigator's discretion (except for prohibited medications: during the treatment period with IV zanamivir, other influenza antiviral drugs were not permitted). The number of participants who were treated with antibiotics for influenza complications was summarized.
Time Frame: Up to post-treatment (PT) + 23 days
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14
Participants | 63 | 5 | 7 | 7 | 12 | 6

29. Secondary Outcome: Median Duration of Hospitalization and Intensive Care Unit (ICU) Stays
Description: The duration of hospitalization (H) reflects the number of hospitalization days between the date of the first dose of investigational product and the date of discharge. ICU stay includes total duration in ICU and may include days in ICU before entry into the study. For participants with a missing discharge date who were not discharged at the end of the study, the date of discharge was imputed to the last follow-up visit (post-treatment +23 days). Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to discharge from hospital
Population: ITT-E Population
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 11 | 12 | 27 | 14
Days
  Duration of H, n=130, 7, 11, 12, 27, 14 | 15.0 [1 to 133] | 7.0 [2 to 23] | 4.0 [2 to 44] | 6.5 [3 to 37] | 6.0 [1 to 45] | 6.5 [2 to 42]
  Duration of H-ICU, n=108, 4, 6, 8, 19, 9 | 11.50 [1 to 104] | 7.5 [5 to 24] | 5.0 [3 to 19] | 5.5 [2 to 26] | 8.0 [2 to 50] | 8.0 [4 to 39]

30. Secondary Outcome: Geometric Mean Maximum Serum Concentration (Cmax) of Zanamivir at the End of Infusion
Description: The Cmax of zanamivir was evaluated at the end of infusion. Serial blood samples for pharmacokinetic (PK) analysis were collected if possible in conjunction with the initial dose on Day 1 (5-7 serial samples) and over a dosing interval during repeat dosing on Days 3, 4, or 5 (5 serial samples). PK data for all participants with available blood samples were analyzed. PK data for those participants who were neither on extracorporeal membrane oxygenation (ECMO) nor on continuous renal replacement therapy (CRRT), who were with CLcr >=80 mL/minutes (>=80mL/minute/1.73m^2 for cohorts 1-4) and who received an initial dose (ID) and a maintenance dose (MD) of 14 mg/kg (6 months to <6 years of age), 12 mg/kg, not to exceed 600 mg (6 to <18 years of age) or 600 mg zanamivir (>=18 years of age) (represented by n=X in the category titles) were summarized. "NA" indicates that data are not available/analysis was not performed.
Time Frame: Day 1 and Days 3, 4, or 5
Population: PK Parameter Population: participants with one or more estimated zanamivir PK parameters
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per mL
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 6 | 12 | 15 | 13
Micrograms per mL
  ID, 600 mg, CLcr>=80, n=67, 0, 0, 0, 0, 6 | 32.77 (34) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 34.47 (27)
  ID, 12 mg/kg, CLcr>=80, n=0, 0, 0, 0, 9, 3 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 44.16 (47) | 4.99 (3997)
  ID, 14 mg/kg, CLcr>=80, n=0, 4, 5, 9, 0, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 36.21 (21) | 37.78 (24) | 41.54 (23) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  MD, 600 mg, CLcr>=80, n=72, 0, 0, 0, 0, 2 | 35.30 (32) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 25.73 (52)
  MD, 12 mg/kg, CLcr>=80, n=0, 0, 0, 0, 4, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 45.18 (48) | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  MD, 14 mg/kg, CLcr>=80, n=0, 0, 1, 4, 0, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 38.01 (NA) — "NA" indicates that data are not available/analysis was not performed. | 43.19 (9) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.

31. Secondary Outcome: Geometric Mean Area Under the Serum Drug Concentration-time Curve (AUC) Over a 12-hour Dosing Interval (AUC[0-tau]) and AUC Extrapolated to Infinity (AUC[0-inf]) of Zanamivir
Description: The AUC(0-tau) during the repeat dose interval and AUC(0-inf) for the initial dose were evaluated. Serial blood samples for PK analysis were collected if possible in conjunction with the initial dose on Day 1 (5-7 serial samples) and over a dosing interval during repeat dosing on Days 3, 4, or 5 (5 serial samples). PK data for all participants with available blood samples were analyzed. PK data for those participants with a CLcr >=80 mL/minutes (>=80 mL/minute/1.73m^2 for cohorts 1-4) and who received an ID and a MD of 14 mg/kg (6 months to <6 years of age), 12 mg/kg, not to exceed 600 mg (6 to <18 years of age) or 600 mg zanamivir (>=18 years of age) (represented by n=X in the category titles) were summarized. "NA" indicates that data are not available/analysis was not performed.
Time Frame: Day 1 and Days 3, 4, or 5
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms*hour per milliliter
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 6 | 12 | 15 | 13
Micrograms*hour per milliliter
  AUC(0-inf), ID, 600 mg, CLcr>=80, n=63,0,0,0,0,5 | 82.86 (36) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 91.07 (27)
  AUC(0-inf), ID, 12 mg/kg, CLcr>=80, n=0,0,0,0,8,1 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 107.21 (41) | 135.22 (NA) — "NA" indicates that data are not available/analysis was not performed.
  AUC(0-inf), ID, 14 mg/kg, CLcr>=80, n=0,3,4,9,0,0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 75.31 (23) | 72.42 (14) | 80.28 (38) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  AUC(0-tau), MD, 600 mg, CLcr>=80, n=65,0,0, 0,0,2 | 90.33 (36) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 64.52 (30)
  AUC(0-tau), MD, 12 mg/kg, CLcr>=80, n=0,0,0,0,4,0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 90.33 (45) | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  AUC(0-tau), MD, 14 mg/kg, CLcr>=80, n=0,0,1,4,0,0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 68.20 (NA) — "NA" indicates that data are not available/analysis was not performed. | 81.02 (28) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.

32. Secondary Outcome: Geometric Mean Terminal Half Life (t1/2) of Zanamivir
Description: The t1/2 of zanamivir was evaluated. Terminal half life is defined as the time it takes for a substance to lose half of its pharmacologic, physiologic, or radiologic activity. Serial blood samples for PK analysis were collected if possible in conjunction with the initial dose on Day 1 (5-7 serial samples) and over a dosing interval during repeat dosing on Day 3, 4, or 5 (5 serial samples). PK data for all participants with available blood samples were analyzed. PK data for those participants with a CLcr>=80 mL/minutes (>=80 mL/minute/1.73m^2 for cohorts 1-4) and who received an ID and a MD of 14 mg/kg (6 months to <6 years of age), 12 mg/kg, not to exceed 600 mg (6 to <18 years of age) or 600 mg zanamivir (>=18 years of age) (represented by n=X in the category titles) were summarized. "NA" indicates that data are not available/analysis was not performed.
Time Frame: Day 1 and Days 3, 4, or 5
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 6 | 12 | 15 | 13
Hours
  ID, 600 mg, CLcr>=80, n=67, 0, 0, 0, 0, 5 | 2.39 (31) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 2.06 (47)
  ID, 12 mg/kg, CLcr>=80, n=0, 0, 0, 0, 8, 1 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 2.57 (55) | 2.16 (NA) — "NA" indicates that data are not available/analysis was not performed.
  ID, 14 mg/kg, CLcr>=80, n=0, 3, 5, 9, 0, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 1.84 (19) | 2.49 (118) | 1.60 (34) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  MD, 600 mg, CLcr>=80, n=68, 0, 0, 0, 0, 2 | 2.56 (34) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 1.73 (21)
  MD, 12 mg/kg, CLcr>=80, n=0, 0, 0, 0, 4, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 1.81 (41) | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  MD, 14 mg/kg, CLcr>=80, n=0, 0, 1, 4, 0, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 1.68 (NA) — "NA" indicates that data are not available/analysis was not performed. | 1.76 (20) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.

33. Secondary Outcome: Geometric Mean Serum Clearance of Zanamivir
Description: The serum clearance of zanamivir was evaluated. Clearance is defined as the volume of zanamivir per unit time eliminated from serum. Serial blood samples for PK analysis were collected if possible in conjunction with the initial dose on Day 1 (5-7 serial samples) and over a dosing interval during repeat dosing on Days 3, 4, or 5 (5 serial samples). PK data for all participants with available blood samples were analyzed. PK data for those participants with a CLcr >=80 mL/minutes (>=80 mL/minute/1.73m^2 for cohorts 1-4) and who received an ID and a MD 14 mg/kg (6 months to <6 years of age), 12 mg/kg, not to exceed 600 mg (6 to <18 years of age) or 600 mg zanamivir (>=18 years of age) (represented by n=X in the category titles) were summarized. "NA" indicates that data are not available/analysis was not performed.
Time Frame: Day 1 and Days 3, 4, or 5
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL per minutes
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 6 | 12 | 15 | 13
mL per minutes
  ID, 600 mg, CLcr>=80, n=63, 0, 0, 0, 0, 5 | 120.68 (36) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 109.83 (27)
  ID, 12 mg/kg, CLcr>=80, n=0, 0, 0, 0, 8, 1 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 46.70 (47) | 53.70 (NA) — "NA" indicates that data are not available/analysis was not performed.
  ID, 14 mg/kg, CLcr>=80, n=0, 3, 4, 9, 0, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 27.31 (32) | 31.00 (12) | 41.95 (37) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  MD, 600 mg, CLcr>=80, n=65, 0, 0, 0, 0, 0 | 110.71 (36) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 155.03 (30)
  MD, 12 mg/kg, CLcr>=80, n=0, 0, 0, 0, 4, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 68.61 (34) | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  MD, 14 mg/kg, CLcr>=80, n=0, 0, 1, 4, 0, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 31.78 (NA) — "NA" indicates that data are not available/analysis was not performed. | 40.35 (35) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.

34. Secondary Outcome: Geometric Mean Volume of Distribution (Vd) of Zanamivir
Description: The Vd of zanamivir was evaluated. Volume of distribution is defined as the apparent volume in which zanamivir is distributed. Serial blood samples for PK analysis were collected if possible in conjunction with the initial dose on Day 1 (5-7 serial samples) and over a dosing interval during repeat dosing on Days 3, 4, or 5 (5 serial samples). PK data for all participants with available blood samples were analyzed. PK data for those participants with a CLcr >= 80 mL/minutes (>=80 mL/minute/1.73m^2 for cohorts 1-4) and who received an ID and a MD of 14 mg/kg (6 months to <6 years of age), 12 mg/kg, not to exceed 600 mg (6 to <18 years of age) or 600 mg zanamivir (>=18 years of age) (represented by n=X in the category titles) were summarized. "NA" indicates that data are not available/analysis was not performed.
Time Frame: Day 1 and Days 3, 4, or 5
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Number analyzed (Participants) | 130 | 7 | 6 | 12 | 15 | 13
Liters (L)
  ID, 600 mg, CLcr>=80, n=63, 0, 0, 0, 0, 5 | 24.89 (27) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 18.57 (26)
  ID, 12 mg/kg, CLcr>=80, n=0, 0, 0, 0, 8, 1 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 9.21 (48) | 10.09 (NA) — "NA" indicates that data are not available/analysis was not performed.
  ID, 14 mg/kg, CLcr>=80, n=0, 3, 4, 9, 0, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 3.77 (12) | 3.94 (29) | 5.15 (20) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  MD, 600 mg, CLcr>=80, n=65, 0, 0, 0, 0, 0 | 24.61 (32) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 23.20 (25)
  MD, 12 mg/kg, CLcr>=80, n=0, 0, 0, 0, 8, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 9.82 (8) | NA (NA) — "NA" indicates that data are not available/analysis was not performed.
  MD, 14 mg/kg, CLcr>=80, n=0, 0, 1, 4, 0, 0 | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | 3.77 (NA) — "NA" indicates that data are not available/analysis was not performed. | 5.23 (32) | NA (NA) — "NA" indicates that data are not available/analysis was not performed. | NA (NA) — "NA" indicates that data are not available/analysis was not performed.

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs) were collected from the start of study medication until follow-up (up to 33 days). Serious adverse events (SAEs) assessed as related to study participation were recorded from time of consent until any follow up contact.
Arm/Group | Cohort 6: Adults (18 Years and Older) | Cohort 1: Infants (6 Months to <1 Year of Age) | Cohort 2: Children (1 to <2 Years of Age) | Cohort 3: Children (2 to <6 Years of Age) | Cohort 4: Children (6 to <13 Years of Age) | Cohort 5: Adolescents (13 to <18 Years of Age)
Serious Adverse Events (participants affected / at risk) | 44/130 | 1/7 | 2/11 | 0/12 | 8/27 | 4/14
Other Adverse Events (participants affected / at risk) | 100/130 | 4/7 | 7/11 | 8/12 | 20/27 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 6: Adults (18 Years and Older) (N=130) | Cohort 1: Infants (6 Months to <1 Year of Age) (N=7) | Cohort 2: Children (1 to <2 Years of Age) (N=11) | Cohort 3: Children (2 to <6 Years of Age) (N=12) | Cohort 4: Children (6 to <13 Years of Age) (N=27) | Cohort 5: Adolescents (13 to <18 Years of Age) (N=14)
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 3 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 4 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 3 | 0 | 0 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 7 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral pericarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 6: Adults (18 Years and Older) (N=130) | Cohort 1: Infants (6 Months to <1 Year of Age) (N=7) | Cohort 2: Children (1 to <2 Years of Age) (N=11) | Cohort 3: Children (2 to <6 Years of Age) (N=12) | Cohort 4: Children (6 to <13 Years of Age) (N=27) | Cohort 5: Adolescents (13 to <18 Years of Age) (N=14)
Hypotension (Vascular disorders) | 15 | 0 | 1 | 0 | 2 | 0
Hypertension (Vascular disorders) | 11 | 0 | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 2 | 0 | 0
Thrombophlebitis (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoperfusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 14 | 1 | 0 | 1 | 4 | 1
Oedema (General disorders) | 7 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 3 | 0 | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis in device (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Unintentional medical device removal (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 12 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Conduct disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug dependence (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Perineal rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 11 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0 | 0 | 0 | 1 | 0
Blood creatinine phosphokinase increased (Investigations) | 2 | 0 | 1 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyl transferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gastric occult blood positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Haematrocrit decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Occult blood positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Pseudomonas test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dilatation ventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Right atrial dilatation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 11 | 0 | 1 | 0 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bandaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphpenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 0 | 1 | 0
Critical illness polyneuropathy (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Neuromyopathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness exertional (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Keratopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pupillary disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 10 | 0 | 1 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 6 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Impaired gastic emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 0 | 0 | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 1 | 0 | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 4 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 3 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 1 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myositis ossificans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 1 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 1 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Penile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pseudomonas bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Two participants who withdrew consent prior to receiving intravenous zanamivir have not been captured in any of the tables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.